CLINICAL TRIAL: NCT06061289
Title: Effects of Standard Process's SP Detox Balance Dietary Supplements on Metabolic Detoxification
Brief Title: Guided Metabolic Detox Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Standard Process Inc. (Industry)
Collaborators: Northwestern Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SP-016
Record Dates: First submitted 2023-03-10; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Detoxification Response
Keywords: Detoxification; Whole Food Vitamins; Glutathione; liver; antioxidants; SOD; GST

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education and healthy diet (No Intervention): The healthy diet education session included a PowerPoint presentation on healthy dietary guidelines and sample recipes of healthy meals.
- Detox (Experimental): The guided component of the detoxification program included an additional PowerPoint presentation with the information about the investigational product, directions, and dosing information for its consumption.
  Interventions: Dietary Supplement: SP Detox Program

INTERVENTIONS:
Dietary Supplement: SP Detox Program — The production use and disposal of toxic chemicals and synthetic materials have increased the risk of exposure to health-threatening toxins. Causal relationships between toxic chemicals and diseases have been well established. However, many patients endure chronic symptoms that are associated with exposure to toxins before advanced stages of specific diseases are realized. Thus, there is a great demand for noninvasive laboratory tests that can provide timely assessment of chemical exposure and the capability of hepatic detoxification
  Arms: Detox

SUMMARY:
Adequate antioxidant supply is essential for maintaining metabolic homeostasis and reducing oxidative stress during detoxification. The emerging evidence suggests that certain classes of phytonutrients can help support the detoxification process by stimulating the liver to produce detoxification enzymes or acting as antioxidants that neutralize the harmful effects of free radicals. This study was designed to examine the effects of a guided 28-day metabolic detoxification program in healthy adults. The participants were randomly assigned to consume a whole food, multi-ingredient supplement (education and intervention) or control (education and healthy meal) daily for the duration of the trial.

DETAILED DESCRIPTION:
In this study, the focus is on a cohort of healthy adults enrolled in a guided detoxification program that included a healthy diet education session with or without 28-day nutritional supplementation with a whole food, proprietary multicomponent blend. The primary objective was to determine the improvement in quality of life by a validated self-reported wellness questionnaire known as Promis Global 10. The secondary outcomes were to quantify the functional markers of metabolic detoxification in blood and urine compared to the study baseline to understand the efficacy of the study formulation as part of 28-day nutritional supplementation with a whole food, proprietary multicomponent blend.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to comply with study protocol for 30 days
* No allergy to any study products (check formulation section below)
* Participant is over 18 years of age or older
* Participant is a male or a non-pregnant, non-lactating female, at least 6 weeks postpartum prior to screening visit, and is not actively planning a pregnancy.
* Participant has at least two weeks wash out period between completion of a previous research study that required ingestion of any study food or drug and their start in the current study.

Exclusion Criteria:

* Prohibited Medications, Supplements or Herbal Products

  * Subjects who are experiencing any adverse events due to any nutraceutical, OTC, or pharmaceutical or investigational products
  * Celiac and other gastrointestinal health concerns
  * Subjects may not receive any other investigational products not part of normal clinical care
  * Lipid lowering drugs or the use of anticoagulant medications in the preceding 4 weeks and for duration of study
* Pregnant and nursing women are excluded from participation and women of childbearing age expecting to be pregnant soon will be excluded from the study
* TC levels less than 220
* Subjects with untreated endocrine, neurological, or infectious disease
* Subjects with the diagnosis of HIV disease or AIDS
* Significant liver or kidney disease (recent or ongoing hepatitis, cirrhosis, glomerulonephritis, dialysis treatment)
* Rheumatoid arthritis, ankylosing spondylitis, systemic lupus erythematosus, polymyositis, scleroderma, polymyalgia rheumatic, temporal arteritis or Reiter's Syndrome
* Psoriasis, Deep vein thrombosis or pulmonary embolus (blood clot to lungs)
* History of cancer
* Serious medical illness
* Substance Use - Use of ethanol within 24 hours of the evaluation visits (baseline, 4 weeks)
* Any other sound medical, psychiatric and/or social reason as determined by the PI
* Co-enrollment in other studies is restricted. Study staff should be notified of co-enrollment as it may require the approval of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-03-06 (Actual); Primary Completion 2022-08-27 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Promis Global 10 (Self- reported Wellness) Questionnaire | 28 days
  The PROMIS Global short form was scored into a Global Physical Health component and Global Mental Health component. The summed raw scores from PROMIS Global were converted into standardized T-score distributions such that a 50 represents the average (mean) for the US general population. A high score always represents more of the concept being measured.

SECONDARY OUTCOMES:
Total Serum Antioxidants | 28 days
  Total Antioxidant Capacity ( μM ) measured as the combined antioxidant activities of all serum constituents, including vitamins, proteins, lipids, glutathione, and uric acid. This assay will be performed using a commercial kit following manufacturer's instruction.
Oxidative Stress | 28 days
  Colorimetric method to study redox status of peripheral blood mononuclear cells (PBMCs) in Relative fluorescence units (RFU)
Detoxification Enzyme Activity - SOD | 28 days
  Assessment of SOD activity (units/mL) using an assay that utilizes a tetrazolium salt for detection of superoxide radicals generated by xanthine oxidase and hypoxanthine using a colorimetric method.
Detoxification Enzyme Activity - GST | 28 days
  Total GST activity (units/mL) measured by quantifying the conjugation of 1-chloro-2,4-dinitrobenzene (CDNB) with reduced glutathione using a glutathione S-transferase assay kit
Urinary Detox marker | 28 days
  Excreted Porphyrins concentration in urine (nmol/mg)
Hepatic detox marker -1 | 28 days
  Excreted D-glucaric acid concentration in urine ((nM/mg)
Hepatic detox marker -2 | 28 days
  Excreted Mercapturic acid concentration in urine ((μM/mM)
Total Glutathione | 28 days
  Serum concentration of Glutathione (uM) was measured as part of a fluorometric assay.

CONTACTS AND LOCATIONS:
Overall Officials: Chinmayee Panda, PhD, Principal Investigator — Standard Process Inc.
Locations (1):
- De-Rusha Clinic, Northwestern Health Sciences University, Bloomington, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sears ME, Genuis SJ. Environmental determinants of chronic disease and medical approaches: recognition, avoidance, supportive therapy, and detoxification. J Environ Public Health. 2012;2012:356798. doi: 10.1155/2012/356798. Epub 2012 Jan 19. PMID 22315626
- [Background] Bonakdar RA, Sweeney M, Dalhoumi S, Adair V, Garvey C, Hodge T, Herrala L, Barbee A, Case C, Kearney J, Smith K, Hwang J. Detoxification Enhanced Lifestyle Intervention Targeting Endotoxemia (DELITE) in the Setting of Obesity and Pain: Results of a Pilot Group Intervention. Integr Med (Encinitas). 2020 Oct;19(5):16-28. PMID 33488302
- [Background] Mostafalou S, Abdollahi M. Pesticides and human chronic diseases: evidences, mechanisms, and perspectives. Toxicol Appl Pharmacol. 2013 Apr 15;268(2):157-77. doi: 10.1016/j.taap.2013.01.025. Epub 2013 Feb 9. PMID 23402800
- [Background] Jochmanova I, Lazurova Z, Rudnay M, Bacova I, Marekova M, Lazurova I. Environmental estrogen bisphenol A and autoimmunity. Lupus. 2015 Apr;24(4-5):392-9. doi: 10.1177/0961203314560205. PMID 25801882
- [Background] Liska D, Lyon M, Jones DS. Detoxification and biotransformational imbalances. Explore (NY). 2006 Mar;2(2):122-40. doi: 10.1016/j.explore.2005.12.009. No abstract available. PMID 16781626
- [Background] Polanska K, Jurewicz J, Hanke W. Review of current evidence on the impact of pesticides, polychlorinated biphenyls and selected metals on attention deficit / hyperactivity disorder in children. Int J Occup Med Environ Health. 2013 Mar;26(1):16-38. doi: 10.2478/s13382-013-0073-7. Epub 2013 Mar 22. PMID 23526196
- [Background] Hodges RE, Minich DM. Modulation of Metabolic Detoxification Pathways Using Foods and Food-Derived Components: A Scientific Review with Clinical Application. J Nutr Metab. 2015;2015:760689. doi: 10.1155/2015/760689. Epub 2015 Jun 16. PMID 26167297
- [Background] Proudfoot AT, Krenzelok EP, Vale JA. Position Paper on urine alkalinization. J Toxicol Clin Toxicol. 2004;42(1):1-26. doi: 10.1081/clt-120028740. PMID 15083932
- [Background] Berardi JM, Logan AC, Rao AV. Plant based dietary supplement increases urinary pH. J Int Soc Sports Nutr. 2008 Nov 6;5:20. doi: 10.1186/1550-2783-5-20. PMID 18990209
- [Background] Konig D, Muser K, Dickhuth HH, Berg A, Deibert P. Effect of a supplement rich in alkaline minerals on acid-base balance in humans. Nutr J. 2009 Jun 10;8:23. doi: 10.1186/1475-2891-8-23. PMID 19515242
- [Background] Minich DM, Bland JS. Acid-alkaline balance: role in chronic disease and detoxification. Altern Ther Health Med. 2007 Jul-Aug;13(4):62-5. PMID 17658124
- [Background] Griendling KK, Touyz RM, Zweier JL, Dikalov S, Chilian W, Chen YR, Harrison DG, Bhatnagar A; American Heart Association Council on Basic Cardiovascular Sciences. Measurement of Reactive Oxygen Species, Reactive Nitrogen Species, and Redox-Dependent Signaling in the Cardiovascular System: A Scientific Statement From the American Heart Association. Circ Res. 2016 Aug 19;119(5):e39-75. doi: 10.1161/RES.0000000000000110. Epub 2016 Jul 14. PMID 27418630
- [Background] Zweier JL, Duke SS, Kuppusamy P, Sylvester JT, Gabrielson EW. Electron paramagnetic resonance evidence that cellular oxygen toxicity is caused by the generation of superoxide and hydroxyl free radicals. FEBS Lett. 1989 Jul 31;252(1-2):12-6. doi: 10.1016/0014-5793(89)80881-6. PMID 2547649
- [Background] Pastore A, Federici G, Bertini E, Piemonte F. Analysis of glutathione: implication in redox and detoxification. Clin Chim Acta. 2003 Jul 1;333(1):19-39. doi: 10.1016/s0009-8981(03)00200-6. PMID 12809732
- [Background] Lee DH, Blomhoff R, Jacobs DR Jr. Is serum gamma glutamyltransferase a marker of oxidative stress? Free Radic Res. 2004 Jun;38(6):535-9. doi: 10.1080/10715760410001694026. PMID 15346644
- [Background] Chen CA, Wang TY, Varadharaj S, Reyes LA, Hemann C, Talukder MA, Chen YR, Druhan LJ, Zweier JL. S-glutathionylation uncouples eNOS and regulates its cellular and vascular function. Nature. 2010 Dec 23;468(7327):1115-8. doi: 10.1038/nature09599. PMID 21179168
- [Background] Varadharaj S, Kelly OJ, Khayat RN, Kumar PS, Ahmed N, Zweier JL. Role of Dietary Antioxidants in the Preservation of Vascular Function and the Modulation of Health and Disease. Front Cardiovasc Med. 2017 Nov 1;4:64. doi: 10.3389/fcvm.2017.00064. eCollection 2017. PMID 29164133
- [Background] Yen CH, Tseng YH, Kuo YW, Lee MC, Chen HL. Long-term supplementation of isomalto-oligosaccharides improved colonic microflora profile, bowel function, and blood cholesterol levels in constipated elderly people--a placebo-controlled, diet-controlled trial. Nutrition. 2011 Apr;27(4):445-50. doi: 10.1016/j.nut.2010.05.012. Epub 2010 Jul 10. PMID 20624673
- [Background] Chen HL, Lu YH, Lin JJ, Ko LY. Effects of isomalto-oligosaccharides on bowel functions and indicators of nutritional status in constipated elderly men. J Am Coll Nutr. 2001 Feb;20(1):44-9. doi: 10.1080/07315724.2001.10719013. PMID 11294172
- [Background] Zhao ZY, Liang L, Fan X, Yu Z, Hotchkiss AT, Wilk BJ, Eliaz I. The role of modified citrus pectin as an effective chelator of lead in children hospitalized with toxic lead levels. Altern Ther Health Med. 2008 Jul-Aug;14(4):34-8. PMID 18616067
- [Background] Zhang N, Huang C, Ou S. In vitro binding capacities of three dietary fibers and their mixture for four toxic elements, cholesterol, and bile acid. J Hazard Mater. 2011 Feb 15;186(1):236-9. doi: 10.1016/j.jhazmat.2010.10.120. Epub 2010 Nov 9. PMID 21095057
- [Background] Eliaz I, Hotchkiss AT, Fishman ML, Rode D. The effect of modified citrus pectin on urinary excretion of toxic elements. Phytother Res. 2006 Oct;20(10):859-64. doi: 10.1002/ptr.1953. PMID 16835878
- [Background] Cuervo A, Salazar N, Ruas-Madiedo P, Gueimonde M, Gonzalez S. Fiber from a regular diet is directly associated with fecal short-chain fatty acid concentrations in the elderly. Nutr Res. 2013 Oct;33(10):811-6. doi: 10.1016/j.nutres.2013.05.016. Epub 2013 Jul 26. PMID 24074739
- [Background] Cline JC. Nutritional aspects of detoxification in clinical practice. Altern Ther Health Med. 2015 May-Jun;21(3):54-62. PMID 26026145
- See also: Urine pH test — https://www.nlm.nih.gov/medlineplus/ency/article/003583.htm